CLINICAL TRIAL: NCT05758961
Title: Le French Gut : the French Microbiota
Brief Title: Le French Gut: Characterization of Gut Microbiota Profiles in France
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Assistance Publique Hopitaux de Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-A01439-32
Record Dates: First submitted 2023-02-01; First posted 2023-03-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: General Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
" The French Gut " is a national contribution aiming to collect 100,000 faecal samples and associated nutritional and clinical data by 2027. Le French Gut is initiated by MetaGenoPolis-INRAE, supported by INRAE with Prof. R. Benamouzig, (AP-HP) as principal investigator of the project. The main goal of this national trial is a better understanding of the observed heterogeneity between gut microbiome of healthy subjects, its connections with the diet and lifestyle, but also changes in gut microbiota associated with diseases (diabetes, obesity, allergies, cancer, Parkinson, Alzheimer…).

DETAILED DESCRIPTION:
At the 14th International Conference on Genomics (ICG-14), scientists from China, Sweden, Denmark, France and Latvia launched The Million Microbiome of Humans Project (MMHP) and agreed to collaborate on a large-scale microbial metagenomic project. The overarching goal is to build the world's largest database of human microbiota with one million microbial samples from the intestines, mouth, skin and reproductive system. Therefore, making it possible to characterize the microbiota of people according to age, gender, height, weight, etc.

As a founding member of the MMHP, INRAE will bring the French national contribution: 100 000 faecal samples and associated nutritional and clinical data from France, by 2027, through Le French Gut project. Initiated by the MGP research unit, Le French Gut is led by INRAE and the AP-HP (Public Assistance-Hospitals of Paris), with the support and collaboration of a consortium of members from medical, scientific and industrial sectors.

In order to be a participant of the project, volunteers will need to fill out an online questionnaire with 60 questions about their lifestyle, their dietary habits and their medical background. The second requirement is the stool sampling, at home.

Main scientific targets of this project are the following:

* Build a map of the intestinal microbiota in France, reflecting differences in term of gut microbiome through ages, gender, regions of life, diets, habits and medical status;
* Describe and better understand the heterogeneity between gut microbiota of healthy subjects and investigate the connection between this heterogeneity with diet and habits.
* Describe the variations of the intestinal microbiota associated with the presence and development of certain diseases (chronic diseases, neurodevelopmental disorders, neurodegenerative diseases,…)

ELIGIBILITY:
Inclusion Criteria:

* Persons over the age of 18 living in France.
* Consent form signed electronically.

Non inclusion Criteria:

* Non-adult person (declarative);
* Person not living in France (declarative);
* Persons subject to a protective measure, in particular under guardianship or curatorship or unable to express their consent (declarative);
* Person having had a colectomy (declarative);
* Person with a digestive stoma (declarative);
* Person who has not signed the consent;
* Person who did not answer the entry questionnaire;
* Person who has not sent a compliant stool sample;
* Antibiotic intake in the 3 months before inclusion (declarative);
* Performing a colonoscopy in the 3 months preceding inclusion (declarative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population residing in France
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2042-09-15 (Estimated)

PRIMARY OUTCOMES:
Characterize the heterogeneity and diversity of the gut microbiota of subjects living in France | 5 up to 15 years
  The gut microbiota of participants will be characterized by describing the presence and abundance in the samples of each gut microbial genes listed in our up-to-date gene catalogue. From these data, the presence and abundance of the different taxonomic ranks will be deduced, ranging from a fine granularity at species and strain level to a more 'zoomed out' phylum level. The richness and diversity of the microbiome (genes and species) will be described. The functional modules, corresponding to the metabolic pathways encoded by the species detected in each sample, will be determined.

SECONDARY OUTCOMES:
Study the variations in the gut microbiota as a function of microbial profile | 5 up to 15 years
Study the variations in the gut microbiota as a function of age | 5 up to 15 years
Study the variations in the gut microbiota as a function of socio-demographic and anthropometric characteristics | 5 up to 15 years
  Richness and diversity of the microbiota (genes and species);
Study the variations in the gut microbiota as a function of lifestyle and eating habits | 5 up to 15 years
Study the variations in the gut microbiota as a function of presence of known pathologies at inclusion, occurrence during follow-up of certain pathologies identified by analysis of data from health from health questionnaires and SNDS data. | 5 up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, Pr, Principal Investigator — APHP; Joël DORE, Pr, Study Chair — INRAE
Locations (1):
- Centre de Recherche sur Volontaire, Bobigny, France

REFERENCES:
- [Derived] Connan C, Fromentin S, Benallaoua M, Alvarez AS, Pons N, Quinquis B, Morabito C, Nazare JA, Borezee-Durant E; Le French Gut Consortium; Haimet F, Ehrlich SD, Valeille K, Cavezza A, Blottiere H, Veiga P, Almeida M, Dore J, Benamouzig R. Associations Among Diet, Health, Lifestyle, and Gut Microbiota Composition in the General French Population: Protocol for the Le French Gut - Le Microbiote Francais Study. JMIR Res Protoc. 2025 May 13;14:e64894. doi: 10.2196/64894. PMID 40358997